CLINICAL TRIAL: NCT02237898
Title: SCH: INT: Harnessing the Power of Technology: MOMBA for Postpartum Smoking
Brief Title: Harnessing the Power of Technology: MOMBA for Postpartum Smoking
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1407014326; 5R01CA195654 (NIH)
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Smoking Cessation
Keywords: Tobacco cessation
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MoMba Contingency Management (Experimental): Study will provide access to the web-based MoMba Live Long application & Sensodrone™ carbon-monoxide sensor for purposes of researching the acceptability of the smartphone application, operating and functioning of it, and providing remote contingency management for smoking cessation to postpartum women.
  Interventions: Behavioral: MoMba Live Long app & Sensordrone™ carbon-monoxide sensor; Device: Sensordrone™ carbon-monoxide sensor; Device: MoMba Live Long Smartphone application
- Office contingency management (Active Comparator): Traditional contingency management with financial incentives delivered in-person in the office for smoking cessation to postpartum women
  Interventions: Behavioral: Office contingency management; Device: Sensordrone™ carbon-monoxide sensor

INTERVENTIONS:
Behavioral: MoMba Live Long app & Sensordrone™ carbon-monoxide sensor — MoMba Live Long application & Sensordrone™ carbon-monoxide sensor to deliver contingency management remotely
  Arms: MoMba Contingency Management
Behavioral: Office contingency management — A control group which will receive financial incentives at an in-person office/clinic visit based on expired CO levels obtained through the piCO sensor.
  Arms: Office contingency management
Device: Sensordrone™ carbon-monoxide sensor — A custom breath CO meter built by Sensorcon Inc. (Sensordrone, part No. SDRONEG1) that uses an electrochemical CO gas sensor to measure environmental CO. The Sensordrone is accurate to within 10% with a resolution of 1 parts per million (ppm). The Sensordrone pairs via Bluetooth with the MoMba Live Long application.
Device: MoMba Live Long Smartphone application — The MoMba Live Long app provides an interface for the Sensordrone which allows participants to complete a breath test and see results of smoking status. The app verifies the user is correctly taking the tests by recording pictures using the front facing camera as well as recording audio to verify that the participants where exhaling while taking the test. The app also provided a platform for social interaction based on a previous system where app users can interact with each other and provide support during the quitting process.
  Arms: MoMba Contingency Management

SUMMARY:
Through a smartphone platform, financial incentives for smoking abstinence in postpartum women can be delivered remotely, thus minimizing the need for participants to come to the office to receive traditional contingency management.

DETAILED DESCRIPTION:
The specific aims of the proposal are:

1. To develop through a 15-month pilot study, a novel smartphone-based system, Momba Smoking, that can be used in further relapse prevention trials for postpartum smokers.
2. To determine, through a pilot randomized controlled trial, the potential feasibility, acceptability, and methodological parameters that are necessary to design a subsequent, appropriately powered, randomized controlled trial of the Momba Smoking smartphone-based system.
3. To advance discovery and understanding on the use of technology to translate smoking cessation interventions from clinical to community settings through the training of the next generation of scientists.

ELIGIBILITY:
Inclusion Criteria:

* Women who are over the age of 18
* Speak English
* Second or third trimester of pregnancy
* Smoking in the third trimester of pregnancy
* No complicating general medical or psychiatric conditions (including marijuana use).

Exclusion Criteria:

* Receiving other smoking cessation medication
* Planning to move out of New Haven in the next 15 months
* Actively suicidal, psychotic or unable to provide informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan V Smith, DrPH, Principal Investigator — Yale University
Locations (1):
- Center for Wellbeing of Women and Mothers, 40 Temple Street, Ste 6B, Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valencia S, Callinan L, Shic F, Smith M. Evaluation of the MoMba Live Long Remote Smoking Detection System During and After Pregnancy: Development and Usability Study. JMIR Mhealth Uhealth. 2020 Nov 24;8(11):e18809. doi: 10.2196/18809. PMID 33231550

RESULTS

PARTICIPANT FLOW:
Groups:
- MoMba Contingency Management: MoMba Contingency Management arm accesses the web-based MoMba Live Long application & Sensodrone™ to research the acceptability and functionality of the app and provides remote contingency management for smoking cessation.
  The Sensordrone™ carbon-monoxide (CO) sensor is a custom breath CO meter built by Sensorcon Inc. (Sensordrone, part No. SDRONEG1) that uses an electrochemical CO gas sensor to measure environmental CO. The Sensordrone is accurate within 10% with a resolution of 1 parts per million (ppm).
  The MoMba Live Long app provides an interface for the Sensordrone allowing participants to complete a breath test. The app allows for verification of completion of the test through pictures and audio recording. The app also provided a platform for social support during the quitting process.
  Most breath tests will be completed remotely.
- Office Contingency Management: The Office Contingency Management (control) group will receive financial incentives at an in-person office visit based on expired CO levels obtained through the piCO sensor for smoking cessation to postpartum women. Tests will be verified with urine samples and a breath test on the Sensordrone™.
  Sensordrone™ carbon-monoxide sensor: A custom breath CO meter built by Sensorcon Inc. (Sensordrone, part No. SDRONEG1) that uses an electrochemical CO gas sensor to measure environmental CO. The Sensordrone is accurate to within 10% with a resolution of 1 parts per million (ppm). The Sensordrone pairs via Bluetooth with the MoMba Live Long application.
  Control participants will not have access to the MoMba Live Long app.
Period: Overall Study
Arm/Group | MoMba Contingency Management | Office Contingency Management
Started | 12 | 14
Completed 12 Weeks of CM | 7 | 2
Completed 3 Month Follow-up | 6 | 6
Completed 9 Month Follow-up | 6 | 7
Completed 15 Month Follow-up | 8 | 8
Completed | 5 | 2
Not Completed | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MoMba Contingency Management | Office Contingency Management | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.08 (6.17) | 28.93 (5.54) | 29.92 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: White, non-Hispanic | 4 | 3 | 7
  Race / Ethnicity: Black or African American, Non-Hispanic | 4 | 8 | 12
  Race / Ethnicity: White, Hispanic | 1 | 1 | 2
  Race / Ethnicity: Black or African American, Hispanic | 1 | 2 | 3
  Race / Ethnicity: Other | 2 | 0 | 2
Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Score ranging from 0-10, higher score indicates more nicotine dependence.
  units on a scale | 3.58 (2.02) | 4.07 (2.06) | 3.85 (2.01)
Number Cigarettes Per Day in Past Month [Median (Inter-Quartile Range); unit: cigarettes / day] — The question asked to the participant was "How many tobacco cigarettes a day have you smoked on average during the last month?" One measure was collected from this question "the average number of cigarettes smoked per day during the last month" per participant. This "average number of cigarettes smoked per day during the last month" was presented in the description.
  cigarettes / day | 7 [5 to 10] | 7 [4 to 20] | 7 [5 to 10]
Number of cigarettes smoked in past 7 days [Median (Inter-Quartile Range); unit: cigarettes / day] — The number of cigarettes smoked in the past 7 days was collected through the self-report timeline follow-back. The average number of cigarettes smoked per day in the past 7 days was calculated as the sum of number of cigarettes smoked per day divided by 7.
  cigarettes / day | 6 [4.8 to 8.5] | 5.5 [3 to 8] | 6 [4 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: Primary Outcome - Acceptability of the delivery of financial incentives for smoking abstinence in postpartum women through a smartphone platform as compared to traditional, in office contingency management. Acceptability of the smartphone application to low-income, pregnant women defined by the percentage of women who would recommend the site to a friend.
  Question: "How likely is it that you would recommend MoMba LiveLong to a friend who wants to stop smoking?"
Time Frame: 3 and 9 months
Population: This measure was assessed at the 3 and 9 month follow-up assessment. Not all participants who were enrolled completed these assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | MoMba Contingency Management | Office Contingency Management
Number analyzed (Participants) | 6 | 7
Participants
  3 month follow-up assessment: number analyzed (Participants) | 6 | 6
  3 month follow-up assessment: Highly Unlikely | 0 | 0
  3 month follow-up assessment: Unlikely | 1 | 0
  3 month follow-up assessment: Neutral | 0 | 0
  3 month follow-up assessment: Likely | 0 | 2
  3 month follow-up assessment: Highly Likely | 5 | 4
  9-month follow-up assessment: Highly Unlikely | 0 | 0
  9-month follow-up assessment: Unlikely | 0 | 0
  9-month follow-up assessment: Neutral | 1 | 1
  9-month follow-up assessment: Likely | 0 | 2
  9-month follow-up assessment: Highly Likely | 5 | 4

2. Primary Outcome: Enrollment Rate
Description: Primary Outcome - Feasibility of the delivery of financial incentives for smoking abstinence in postpartum women through a smartphone platform as compared to traditional, in office contingency management. Feasibility: participation rate of > 60% for eligible women between screening and enrollment. Number of women who were eligible from screening that completed an intake.
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Groups:
- Eligible From Screening: Women who were eligible for participation in the study from screening.
Arm/Group | Eligible From Screening
Number analyzed (Participants) | 43
Participants | 26

3. Primary Outcome: Remote Detection
Description: Primary outcome is the correlation coefficient. The correlation coefficient was calculated between the piCO+™ and the Sensordrone™ specific to expired CO measurement and verified through urine cotinine levels. Data for all three instruments was collected during week 1 visits 1-5, 3 month, 9 month and 15 month assessments.
Time Frame: 15 months
Population: The correlation between the piCO+™, Sensordrone™ and urine cotinine levels are considered and the unit analyzed is a visit, data collected during the first week of office visits and at follow-up assessments. Of participants enrolled, 4 participants who completed a baseline did not attend week 1 and thus didn't contribute any data to this analysis.
Measure: Number; unit: correlation
Units Other Than Participants: Unique visits
Arm/Group | MoMba Contingency Management | Office Contingency Management
Number analyzed (Participants) | 11 | 11
Number analyzed (Unique visits) | 56 | 53
correlation
  Sensordrone and Pico | 0.93 | 0.87
  Sensordrone and Urine | 0.76 | 0.66
  Pico and Urine | 0.81 | 0.67

4. Primary Outcome: Retention: Number of Participants Remaining in Study at 12 Weeks
Description: Primary Outcome - Feasibility of the delivery of financial incentives for smoking abstinence in postpartum women through a smartphone platform as compared to traditional, in office contingency management. Feasibility: retention set at 80% for the Momba Smoking group. Number of participants in the intervention group (MoMba Contingency Management) and number of participants in the control group (office contingency management) who remained in the study at the end of contingency management (12 weeks).
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | MoMba Contingency Management | Office Contingency Management
Number analyzed (Participants) | 12 | 14
Participants | 7 | 2

5. Primary Outcome: Visit Attendance / Challenge Completion
Description: Primary Outcome - Feasibility of the delivery of financial incentives for smoking abstinence in postpartum women through a smartphone platform as compared to traditional, in office contingency management. Feasibility: challenge completion and in-office visit attendance to assess compliance.
  MoMba Contingency Management: Number of breath tests completed among participants who remained enrolled at the end of 12 weeks.
  Office Contingency Management: Number of breath tests (corresponds to office visits) completed among participants who remained enrolled at the end of 12 weeks.
Time Frame: 15 months
Measure: Median (Inter-Quartile Range); unit: breath tests
Groups:
- MoMba Contingency Management: MoMba Contingency Management arm accesses the web-based MoMba Live Long application & Sensodrone™ to research the acceptability and functionality of the app and provides remote contingency management for smoking cessation.
  The Sensordrone™ carbon-monoxide (CO) sensor is a custom breath CO meter built by Sensorcon Inc. (Sensordrone, part No. SDRONEG1) that uses an electrochemical CO gas sensor to measure environmental CO. The Sensordrone is accurate within 10% with a resolution of 1 parts per million (ppm).
  The MoMba Live Long app provides an interface for the Sensordrone allowing participants to complete a breath test. The app allows for verification of completion of the test through pictures and audio recording. The app also provided a platform for social support during the quitting process..
  Most breath tests will be completed remotely.
Arm/Group | MoMba Contingency Management | Office Contingency Management
Number analyzed (Participants) | 7 | 2
breath tests | 16 [15 to 22] | 21.5 [20 to 23]
Statistical Analysis 1: Comparison: MoMba Contingency Management vs Office Contingency Management; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants With Short Term Abstinence From Smoking
Description: Secondary outcome - Short term abstinence from smoking. Immediate smoking prevalence as determined by # of negative breath tests and self-reports; the pilot will also utilize urine tests to measure negative cotinine levels.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | MoMba Contingency Management | Office Contingency Management
Number analyzed (Participants) | 6 | 6
Participants
  Number of negative breath tests using Sensordrone | 2 | 2
  Number of negative breath tests using piCO | 3 | 2
  Self-report (no smoking cigs in past 7 days) | 3 | 1
  Urine test (<50ng) | 3 | 1

7. Secondary Outcome: Number of Participants With Long Term Abstinence From Smoking at 9 Month Follow-Up
Description: Secondary outcome - Long term abstinence from smoking equals 7-day point prevalence determined through # of negative breath tests and self-reports based on the Timeline Follow Back.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | MoMba Contingency Management | Office Contingency Management
Number analyzed (Participants) | 6 | 7
Participants
  Number of negative breath tests using Sensordrone | 2 | 2
  Number of negative breath tests using the piCO | 3 | 3
  Last 7 days no smoking (from timeline followback) | 1 | 0

8. Secondary Outcome: Number of Participants With Long Term Abstinence From Smoking at 15 Month Follow-Up
Description: as for outcome 7
Time Frame: 15 months
Population: In the intervention group only 7/8 participants had data for the timeline follow back.
Measure: Count of Participants; unit: Participants
Arm/Group | MoMba Contingency Management | Office Contingency Management
Number analyzed (Participants) | 8 | 8
Participants
  Number of negative breath tests using Sensordrone | 3 | 4
  Number of negative breath tests using the piCO | 3 | 4
  Last 7 days no smoking (from timeline followback): number analyzed (Participants) | 7 | 8
  Last 7 days no smoking (from timeline followback) | 1 | 0

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected during the course of the study (enrollment until the last follow-up at 15 months).
Description: The definition does not differ.
  Methods for reporting adverse events: Any serious, unanticipated and related adverse events or unanticipated problems involving risks to subjects or others will be reported in writing within 48 hours to the HIC and any appropriate funding and regulatory agencies. Fellow investigators and study personnel will be informed through regular study meetings and study sponsors will be informed within 5 days of the event becoming known to the principal investigator.
Arm/Group | MoMba Contingency Management | Office Contingency Management
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT02237898/Prot_SAP_000.pdf